CLINICAL TRIAL: NCT00814567
Title: Randomised Trial Testing Intensity Modulated and Partial Organ Radiotherapy After Breast Conservation Surgery for Early Breast Cancer
Brief Title: Radiation Therapy in Women With Low Risk Early-Stage Breast Cancer Who Have Undergone Breast Conservation Surgery
Acronym: IMPORT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: Cancer Research UK (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000629768; NIHR 2253 (Other: NIHR); ICR-CTSU/2006/10001 (Other: ICR-CTSU); ISRCTN12852634 (Registry Identifier: ISRCTN); CRUK/06/003 (Other Grant/Funding Number: Cancer Research UK); 06/Q1605/128 (Other: Main Research Ethics Committee)
Record Dates: First submitted 2008-12-24; First posted 2008-12-25 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer; stage IA breast cancer; stage II breast cancer; invasive ductal breast carcinoma; invasive ductal breast carcinoma with predominant intraductal component
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Ductal, Breast | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm I (control) (Active Comparator): Patients undergo standard whole breast radiotherapy once daily on days 1-5 for 3 weeks.
  Interventions: Radiation: radiation therapy
- Arm II (Experimental): Patients undergo reduced whole breast radiotherapy and standard partial breast radiotherapy once daily on days 1-5 for 3 weeks.
  Interventions: Radiation: radiation therapy
- Arm III (Experimental): Patients undergo standard partial breast radiotherapy once daily on days 1-5 for 3 weeks.
  Interventions: Radiation: radiation therapy

INTERVENTIONS:
Radiation: radiation therapy — Patients undergo standard whole breast, reduced whole breast, or standard partial breast radiotherapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Giving radiation therapy after surgery may kill any tumor cells that remain after surgery. It is not yet known whether intensity-modulated radiation therapy is more effective than standard radiation therapy in treating patients with early-stage breast cancer.

PURPOSE: This randomized phase III trial is comparing radiation therapy regimens in treating women with early-stage breast cancer who have undergone breast-conservation surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* To test partial breast radiotherapy using intensity-modulated techniques following complete local tumor excision in women with low-risk, early stage breast cancer.

OUTLINE: This is a multicenter study.

Patients are stratified according to center (not participating in sub-studies vs participating in sub-studies). Patients are randomized to 1 of 3 treatment arms.

* Arm I (control): Patients undergo standard whole breast radiotherapy once daily on days 1-5 (15 fractions) for 3 weeks.
* Arm II: Patients undergo reduced whole breast radiotherapy (15 fractions) and standard partial breast radiotherapy (15 fractions) once daily on days 1-5 for 3 weeks.
* Arm III: Patients undergo standard partial breast radiotherapy once daily on days 1-5 (15 fractions) for 3 weeks.

All patients complete a family history questionnaire at baseline. Patients also undergo blood sample collection at baseline and paraffin-embedded tissue collection at follow-up for molecular studies analyzing inter-patient variation by microarrays.

Patients in centers participating in sub-studies undergo quality of life and health economic assessment at baseline, 6 months, and 1, 2, and 5 years. These patients also undergo photographic assessment at baseline, 2 years, and 5 years.

After completion of study treatment, patients are followed for 10 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of low-risk early stage breast cancer, meeting the following criteria:

  * Invasive adenocarcinoma

    * No invasive carcinoma of classical lobular type
    * lympho-vascular invasion present or absent
  * Tumor size pathologically determined to be ≤ 3.0 cm in diameter (pT1-2) (< 3.1 cm maximum microscopic diameter of invasive component)
  * Unifocal disease
  * Grade I, II, or III disease
  * Axillary lymph nodes negative or 1-3 nodes positive (pN0 or pN+(1-3))
* Must have undergone breast conservation surgery with or without adjuvant systemic therapy

  * Minimum microscopic margin of non-cancerous tissue ≥ 2 mm (excluding deep margin if this is at deep fascia)
* At low risk of local recurrence after radiotherapy (< 1% annual risk local recurrence)
* No prior mastectomy
* No blood-borne metastases

PATIENT CHARACTERISTICS:

* No prior malignancy except nonmelanoma skin cancer

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior endocrine therapy or chemotherapy

  * Neoadjuvant endocrine therapy allowed provided the tumour is < 3.0 cm and all other inclusion criteria are met
  * No primary endocrine therapy as a replacement for surgery
* No concurrent chemoradiotherapy

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2018 (Actual)
Dates: Start 2007-05-03 (Actual); Primary Completion 2016-06-15 (Actual); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Local tumor control in the ipsilateral breast (i.e., true recurrence plus new primary tumor) as confirmed by cytological or histological assessment | 5 years

SECONDARY OUTCOMES:
Location of tumor relapse | 5 years
Contralateral primary breast cancer or other primary tumors as confirmed by cytological or histological assessment | 5 years
Regional and distant metastases | 5 years
Late adverse effects in normal tissue normal tissues as determined periodically by photographic assessments (in a subset of patients), physician assessments, and patient self-assessments | 5 years
Quality of life as assessed by EORTC QLQ C-30, EORTC QLQ-BR23, BIS, and HADS questionnaires in a subset of patients at baseline, 6 months, and 1, 2, and 5 years | 5 years
Cost-effectiveness as assessed by EQ-5D questionnaire at baseline, 6 months, and 1, 2, and 5 years | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte E Coles, PhD, Principal Investigator — University of Cambrige, England
Locations (1):
- Royal Marsden - Surrey, Sutton, England, United Kingdom

REFERENCES:
- [Background] Coles CE, Griffin CL, Kirby AM, Titley J, Agrawal RK, Alhasso A, Bhattacharya IS, Brunt AM, Ciurlionis L, Chan C, Donovan EM, Emson MA, Harnett AN, Haviland JS, Hopwood P, Jefford ML, Kaggwa R, Sawyer EJ, Syndikus I, Tsang YM, Wheatley DA, Wilcox M, Yarnold JR, Bliss JM; IMPORT Trialists. Partial-breast radiotherapy after breast conservation surgery for patients with early breast cancer (UK IMPORT LOW trial): 5-year results from a multicentre, randomised, controlled, phase 3, non-inferiority trial. Lancet. 2017 Sep 9;390(10099):1048-1060. doi: 10.1016/S0140-6736(17)31145-5. Epub 2017 Aug 2. PMID 28779963
- [Background] Bhattacharya IS, Haviland JS, Kirby AM, Kirwan CC, Hopwood P, Yarnold JR, Bliss JM, Coles CE; IMPORT Trialists. Patient-Reported Outcomes Over 5 Years After Whole- or Partial-Breast Radiotherapy: Longitudinal Analysis of the IMPORT LOW (CRUK/06/003) Phase III Randomized Controlled Trial. J Clin Oncol. 2019 Feb 1;37(4):305-317. doi: 10.1200/JCO.18.00982. Epub 2018 Dec 11. PMID 30532984
- [Background] Kirby AM, Bhattacharya IS, Wilcox M, Haviland JS. The IMPORT LOW Trial: Collaborative Research Accelerates Practice Change in Breast Radiotherapy. Clin Oncol (R Coll Radiol). 2019 Jan;31(1):5-8. doi: 10.1016/j.clon.2018.08.007. Epub 2018 Sep 17. No abstract available. PMID 30236641
- [Background] Coles C, Yarnold J; IMPORT Trials Management Group. The IMPORT trials are launched (September 2006). Clin Oncol (R Coll Radiol). 2006 Oct;18(8):587-90. doi: 10.1016/j.clon.2006.07.010. No abstract available. PMID 17051947